CLINICAL TRIAL: NCT05446909
Title: Modulation Effects of a Novel Body-mind Intervention on Subjective Cognitive Decline
Brief Title: Preventing Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022 IBMT SCD; 3R61AT010138-03S1 (NIH)
Record Dates: First submitted 2022-05-25; First posted 2022-07-07 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: mindfulness vs. health education
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBMT mindfulness (Experimental): An evidence-based preventive intervention - integrative body-mind training (IBMT) has shown positive effects in reducing stress, and improving self-control and brain plasticity related to cognitive performance. It has bodifulness and mindfulness components.
  Interventions: Behavioral: IBMT mindfulness
- health education (Active Comparator): Health education includes health-related topics - exercise, sleep, stress management, nutrition, lifestyle
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: IBMT mindfulness — IBMT is an effortless mindfulness technique; health education is a class including health-related topics - exercise, sleep, nutrition, lifestyle, stress management
  Arms: IBMT mindfulness
Behavioral: health education — Health education includes health-related topics - exercise, sleep, stress management, nutrition, lifestyle
  Arms: health education

SUMMARY:
The study aims to understand the mechanisms and training effects of evidence-based body-mind training on improving cognitive performance and preventing cognitive decline.

DETAILED DESCRIPTION:
Subjective cognitive decline (SCD), the self-reported perception of memory or cognitive problems, is a risk factor for the cognitive decline and development of Alzheimer's (AD) and often happens in midlife. Recently, few mind-body interventions have suggested promising effects in preventing cognitive decline. However, these interventions often require longer training time (months to years) to achieve modest benefits, making them less optimal for rapidly learning and achieving desirable outcomes. One mechanism for cognitive decline and AD may involve deficits in self-control networks, and autonomic nervous system (ANS) and these deficits can be ameliorated through body-mind interventions. This study aims to investigate the modulation effects of a novel body-mind intervention on SCD using an evidence-based preventive intervention - integrative body-mind training (IBMT).

ELIGIBILITY:
Inclusion Criteria:

* Able to read/understand English
* Normal performance using standardized cognitive tests
* Self-reported decline in cognitive capacity such as memory loss
* Eligible for non-invasive fMRI
* Willing to be randomized
* Free of any severe psychiatric diagnoses or medication that may affect participation

Exclusion Criteria:

* Medical disorders or medications that affect the central and autonomic nervous system; or a positive pregnancy test result (females)
* Unable to provide consent or understand study procedures due to mental illness or cognitive limitations
* Previous meditation experiences
* Evidence of illicit drug use
* Participants for blood draws weigh less than 110 lbs
* Metal or metallic materials in the body such as pacemaker

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: YiYuan Tang, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IBMT Mindfulness | Health Education
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IBMT Mindfulness | Health Education | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown/Not Reported Ethnicity | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Trials Correct On Working Memory Test
Description: The percentage of trials correct on N-back working memory test; higher percentage of trials correct mean a better outcome.
Time Frame: The outcome measures are assessed online or/and in-person at baseline and post-intervention (2 weeks).
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 15 | 14
percentage of correct trials
  Baseline | 87.69 (0.15) | 91.57 (0.14)
  Post-Intervention | 88.01 (0.16) | 91.68 (0.17)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p > 0.05, ANOVA

2. Primary Outcome: Intervention Effects on Cognitive Decline
Description: The composite measures of cognition such as subjective cognitive decline; the minimum and maximum values (1 and 27); higher scores mean a worse outcome.
Time Frame: The outcome measures are assessed online or/and in-person at baseline and post-intervention (2 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 15 | 14
score on a scale
  Baseline | 5.34 (1.18) | 4.96 (1.02)
  Post-Intervention | 5.29 (1.17) | 4.87 (1.03)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p > 0.05, ANOVA

3. Primary Outcome: Intervention Effects on Emotion Regulation
Description: The composite measures of executive function such as emotion regulation questionnaire; the minimum and maximum values (4 and 10); higher scores mean a better outcome.
Time Frame: The outcome measures are assessed online or/and in-person at baseline and post-intervention (2 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 15 | 14
score on a scale
  Baseline | 5.71 (0.83) | 5.23 (1.12)
  Post-Intervention | 5.50 (1.21) | 4.94 (0.84)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p > 0.05, ANOVA

4. Primary Outcome: Intervention Effects on Mindfulness
Description: The composite measures of executive function such as Five Facet Mindfulness Questionnaire; the minimum and maximum values (1 and 5); higher scores mean a better outcome.
Time Frame: The outcome measures are assessed online or/and in-person at baseline and post-intervention (2 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 15 | 14
score on a scale
  Baseline | 2.92 (0.29) | 2.87 (0.32)
  Post-Intervention | 3.92 (0.49) | 3.39 (0.50)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p < 0.05, ANOVA

5. Secondary Outcome: Intervention Effects on Brain Function
Description: Changes in the strength of brain functional connectivity were measured by functional resting-state brain imaging. Higher numerical values represent stronger connectivity/better outcomes and lower values represent weaker connectivity/worse outcomes. Arbitrary units are used and the theoretical range of the values is from 0 to 1.
Time Frame: The outcome measures are assessed in-person at baseline and post-intervention (2 weeks).
Population: Only participants who had usable data with good image quality were analyzed and reported.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 10 | 11
arbitrary units
  Baseline | 0.47 (0.31) | 0.51 (0.39)
  Post-intervention | 0.53 (0.33) | 0.49 (0.35)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p = 0.754, ANOVA

6. Secondary Outcome: Intervention Effects on Brain White Matter
Description: Changes in AD-signature cortical brain white matter (i.e., level of fractional anisotropy) were measured by diffusion imaging. Higher numerical values represent higher white matter integrity/better outcomes and lower values represent lower white matter integrity/worse outcomes. Arbitrary units are used and the theoretical range of the values is from 0 to 1.
Time Frame: The outcome measures are assessed in-person at baseline and post-intervention (2 weeks).
Population: Only participants who had usable data with good image quality were analyzed and reported.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 10 | 11
arbitrary units
  Baseline | 0.42 (0.04) | 0.39 (0.05)
  Post-intervention | 0.43 (0.04) | 0.37 (0.04)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p = 0.985, ANOVA

7. Secondary Outcome: Intervention Effects on Brain Grey Matter
Description: Changes in AD-signature cortical grey matter volume were measured by MRI structural imaging. Higher numerical values represent greater grey matter volume/better outcomes and lower values represent lower grey matter volume/worse outcomes.
Time Frame: The outcome measures are assessed in-person at baseline and post-intervention (2 weeks).
Population: Only participants who had usable data with good image quality were analyzed and reported.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | IBMT Mindfulness | Health Education
Number analyzed (Participants) | 10 | 11
cm^3
  Baseline | 589.23 (69.3) | 569.39 (67.32)
  Post-intervention | 570.42 (62.11) | 576.87 (64.28)
Statistical Analysis 1: Comparison: IBMT Mindfulness vs Health Education; Test type: Superiority; p = 0.877, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | IBMT Mindfulness | Health Education
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT05446909/Prot_SAP_ICF_000.pdf